CLINICAL TRIAL: NCT02458066
Title: Cluster Randomised Trial to Compare Effectiveness of Bendiocarb and Deltamethrin (Long-Lasting) in Preventing Malaria Infection
Brief Title: Trial to Compare Effectiveness of 2 Insecticides in Preventing Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Care Development, Inc. (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MedicalCareDev
Record Dates: First submitted 2015-05-13; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — bendiocarb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bendiocarb (Active Comparator): IRS: bendiocarb
  Interventions: Other: IRS: bendiocarb
- Deltamethrin (Active Comparator): IRS: deltamethrin
  Interventions: Other: IRS: deltamethrin

INTERVENTIONS:
Other: IRS: bendiocarb — carbamate insecticide
  Other Names: FICAM
  Arms: Bendiocarb
Other: IRS: deltamethrin — Pyrethroid insecticide
  Other Names: K-Othrine SC 62.5
  Arms: Deltamethrin

SUMMARY:
Twenty-four (24) clusters, each containing between 250-300 houses were selected throughout Bioko Island to be sprayed with either a long lasting pyrethroid insecticide, K-Othrine SC 62.5, or a bendiocarb insecticide, FICAM. Parasite prevalence in children aged 2-14 was measured before and after the application of insecticide.

DETAILED DESCRIPTION:
In 2013, a new long lasting pyrethroid insecticide, K-Othrine SC 62.5, that has been developed by Bayer AG, was used for the IRS program in Bioko Island, Equatorial Guinea, for the first time. This change coincided with a marked increase in parasite prevalence in 2-14 year olds as measured in the Annual Malaria Indicator Survey (14% to 28%, respectively). In order to determine whether the change in insecticide caused the increase in prevalence, a cluster randomized control trial was designed.

Twenty-four (24) clusters, each containing between 250-300 houses were selected throughout Bioko Island. Clusters were chosen with an attempt to maximize the geographical space between clusters (to minimize possible residual effects from insecticides), while ensuring that areas with historically higher acceptance rates for Indoor Residual Spraying (IRS) were selected. Each cluster had a buffer zone of 300m (or halfway between clusters less than 600m apart).

A team of 10 local surveyors conducted a baseline survey in each cluster area, measuring prevalence through malaria Rapid Diagnostic Test (RDT) positivity, net ownership, spray coverage, and hemoglobin levels. Approximately 100 children in each cluster were tested. These data were then used for a restricted randomization. Each cluster was then sprayed with either deltamethrin or bendiocarb, depending on randomization. The IRS team put equal amount of effort into each cluster, as determined by number of sprayers/house/day in an attempt to minimize bias.

An end-line survey was conducted using an ODK Collect application in the same cluster areas. Prevalence was measured by RDT, and hemoglobin data was gathered. In addition, the head of household was asked about the acceptability to IRS and their willingness to receive the insecticide in a future round.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2-14 years old who reside in a household within the intervention area
* Household clusters chosen among those with historically high IRS acceptance rate
* Household clusters chosen to maximize distance between clusters.

Exclusion Criteria:

* Areas with historically high rates of refusing IRS

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2800 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of falciparum infection in 2-14 year olds | 3-5 months post receiving IRS
  Cross sectional Rapid Diagnostic Test (RDT)-based prevalence of infection of P.falciparum in children between the ages of 2 and 14 of the participating localities.

SECONDARY OUTCOMES:
Prevalence of infection, adjusted for potential cofounders in 2-14 year olds | 3-5 months post receiving IRS
  - RDT-based prevalence of infection in children between the ages of 2 and 14 of the participating localities, adjusted for potential confounders, such as bednet use, socio-economic status, age of subjects etc.
Severe anemia in children under 5 | 3-5 months post receiving IRS
  - Severe anaemia prevalence (haemoglobin< 8 g/dL) in children under 5 years of age of the participating localities.